CLINICAL TRIAL: NCT06045338
Title: Mind Body Intervention for Long COVID
Brief Title: Mind Body Intervention for Long COVID-19
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Michael Donnino, Physician, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023P000529
Record Dates: First submitted 2023-09-19; First posted 2023-09-21 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Long COVID; Post-Acute Sequelae of COVID-19; COVID Long-Haul
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mind Body Intervention #1 (Experimental)
  Interventions: Behavioral: Mind Body Intervention #1
- Mind Body Intervention #2 (Active Comparator)
  Interventions: Behavioral: Mind Body Intervention #1
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Mind Body Intervention #1 — The mind-body intervention will include regular 1 to 2 hour educational sessions and lectures, as well as supplemental reading material. In addition, individualized sessions will be offered each week for students who have additional questions and/or need additional time with the material.
  Arms: Mind Body Intervention #1; Mind Body Intervention #2

SUMMARY:
The goal of this study is to determine if a mind-body intervention can help people suffering from symptoms associated with Long COVID. The study is a randomized trial examining the effectiveness of a mind body intervention in reducing somatic symptoms from Long COVID in participants as compared to usual care and an active control (second mind body intervention). The investigators will secondarily investigate whether the intervention alleviates individual somatic complaints and improves daily functioning, relative to usual care and the active control

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥ 18 years of age)
2. Infection with Sars-COV2 (i. e., positive antibody, antigen, or PCR testing)
3. Symptoms attributed only to COVID-19 and not to known comorbid disease (e.g., other infections, cancer, etc)
4. A somatic symptom score ≥ 10 on the SSS-8 questionnaire with involvement of at least 3 domains
5. Symptoms present at least 3 day a week for a minimum of 3 months
6. Willingness to engage in a Mind-Body intervention

Exclusion Criteria:

1. Clear diagnosis of physical disease (e.g. lung fibrosis, myocarditis) not inclusive of non-specific findings such as mild arthritis
2. Hospitalization in an intensive care unit for acute COVID-19 infections
3. Age greater than 65 years
4. Diagnosis of dementia or similar cognitive impairment
5. Active addiction disorder (e.g. cocaine) that would interfere with study participation
6. Major psychiatric comorbidity (e.g., schizophrenia). Mild to moderate anxiety and depression are not considered in this category

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Somatic Symptom Score-8 (SSS-8) | Baseline, 4 weeks, 8 weeks, 13 weeks
  Survey questions pertain to pain, the gastrointestinal system, fatigue, dizziness, and cardiovascular complaints. Range of 0-32, with higher scores indicating higher levels of discomfort.

SECONDARY OUTCOMES:
Short Form Brief Pain Inventory (BPI) | Baseline, 4 weeks, 8 weeks, 13 weeks
  Used to gauge pain intensity, and pain interference with daily function over the duration of the study
Fatigue Severity Scale (FSS) | Baseline, 4 weeks, 8 weeks, 13 weeks
  Consists of statements relating to a patient's general level of fatigue and fatigue with specific activities. Range of 7-63, with higher scores indicating a higher degree of fatigue.
The Multidimensional Dyspnea Profile (MDP) | Baseline, 4 weeks, 8 weeks, 13 weeks
  A survey that assesses perceived physical aspects of dyspnea and associated emotional effects. Each of the rating scales within the MDP is designed to measure a separate construct, though each can be grouped between the two above mentioned domains.
Generalized Anxiety Disorder form 7 (GAD-7) | Baseline and 13 weeks
  Self-report instrument assessing general anxiety over the last two weeks. Each of the 7 item is a statement concerning an anxiety trait, respondents then rate how often that statement is true. Responses range from 0 (not at all) to 3 (nearly every day).
Patient Reported Outcomes Measurement Information System survey for function disability (PROMIS) | Baseline, 4 weeks, 8 weeks, 13 weeks
  a standardized assessment of health-related quality of life
End of study measurements | 13 weeks
  Participants' subjective experience of the program upon completion
Pain Anxiety Symptom Score-20 (Pass-20) | Baseline, 4 weeks, 8 weeks, 13 weeks
  Anxiety from pain determined from 20 item survey, with each item being scored from 1-5 in terms of frequency

CONTACTS AND LOCATIONS:
Overall Officials: Michael Donnino, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No